CLINICAL TRIAL: NCT06424951
Title: Kindness is Lesser Preferable Than Happiness: Investigating Interest in Different Effects of the Loving-kindness and Compassion Meditations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KM202210028001
Record Dates: First submitted 2024-05-14; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Meditation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LKCMs (Experimental)
  Interventions: Behavioral: LKCM(Loving-kindness and Compassion Meditations)

INTERVENTIONS:
Behavioral: LKCM(Loving-kindness and Compassion Meditations) — Loving-kindness and Compassion Meditations

SUMMARY:
As an initial step, Study 1 intended to compare the interest in different effects of LKCM among a convenient sample of university students. In order to separate different effects and close to application in real setting, the study will measure participants' interest in participating in proposed meditations, each of which aimed to generate one specific effect. The kind attitudes were represented by compassion for others, compassion for oneself, and appreciative joy for others, which were emphasized in the real LKCM trainings. The emotional well-being included increasing positive emotion, decreasing negative emotion and improving peacefulness, which were validated effects of LKCM. Other validated effects were also measured as fillers and used as additional explorations. The core hypothesis was that the interest in meditations on kind attitudes is significantly lower than interest in meditations on emotional well-being.

The current study created a measure called Willingness to Participate in Meditation Trainings (WPMT). Participants rated their willingness to participate in nine meditation trainings that serve different purposes. Each meditation was rated by one item ("if the purpose of meditation training is to xxx, how much are you willing to participate?" where "xxx" indicates the purposes listed below) and was measured with a 100-mm Visual Analogue Scale (0 = totally unwilling to participate, 100 = totally willing to participate).

Study 2 adopted WPMT in a 21-day online LKCM training. This make sure all participants really took part in meditation training, and allowed further exploration on how participants' WPMT were associated with the adherence and effects of training. To be more sensitive for the change during short training, the effects of training used state-like measures and still focused on two aspects: (1) personal happiness (happiness, sadness, peacefulness) which matched emotional well-being, and (2) interpersonal relationship (love, hate, gratitude) which reflected kind attitudes. The core hypotheses were that higher interest in meditations on Emotional Well-being and Kind attitudes predicted increases in personal happiness and interpersonal relationship, respectively.

ELIGIBILITY:
For study 1 Participants were recruited from two universities in Mainland China with the help of university staff. No other eligibility tests were required.

For study 2 Participants with or without religious beliefs or meditation experience could participate in the study. Each person is required to complete a 21-day meditation course.

Ages: 16 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1658 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Interest in Different Effects of LKCM Training | 4 months
  The core hypothesis was that the interest in meditations on kind attitudes is significantly lower than interest in meditations on emotional well-being.
  The study created a measure called Willingness to Participate in Meditation Trainings (WPMT). Participants rated their willingness to participate in nine meditation trainings that serve different purposes. Each meditation was rated by one item ("if the purpose of meditation training is to xxx, how much are you willing to participate?" where "xxx" indicates the purposes listed below) and was measured with a 100-mm Visual Analogue Scale (0 = totally unwilling to participate, 100 = totally willing to participate).
Interest in Different Effects and Their Relation with Results of Training | 3 months
  The core hypotheses were that higher interest in meditations on Emotional Well-being and Kind attitudes predicted increases in personal happiness and interpersonal relationship, respectively.
  The study adopted WPMT in a 21-day online LKCM training. The measure of WPMT was basically the same with that in Study 1, and it directly asked the interests in the current 21-day meditation training.
  The measure for effects of training used word lists, which measured the frequency of 10 types of experience in the past week, with three items for each type.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deng Y, Du T, Zeng X, Wang W. Kindness is lesser preferable than happiness: investigating interest in different effects of the loving-kindness and compassion meditations. BMC Psychol. 2025 Apr 26;13(1):443. doi: 10.1186/s40359-025-02771-4. PMID 40287761